CLINICAL TRIAL: NCT00108836
Title: Efficacy, Safety and Tolerability of XBD173 in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXBD173A2204
Record Dates: First submitted 2005-04-19; First posted 2005-04-20 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2007-11

CONDITIONS: Anxiety Disorders
Keywords: GAD; Anxiety; XBD173; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — N-benzyl-N-ethyl-2-(7,8-dihydro-7-methyl-8-oxo-2-phenyl-9H-purin-9-yl)acetamide

INTERVENTIONS:
Drug: XBD173

SUMMARY:
This study will test the efficacy, safety and tolerability of XBD173 in the treatment of generalized anxiety disorder in patients.

ELIGIBILITY:
Inclusion Criteria:

* Current doctor's diagnosis of generalized anxiety disorder
* In need of psychiatric treatment
* Willingness to complete all aspects of the study

Exclusion Criteria:

* Current doctor's diagnosis of major depression
* History of schizophrenia or schizoaffective disorders
* Drug dependence within 2 months prior to study start

For detailed information on eligibility, please contact the study center nearest to you (see below), or call 1-862-778-8300, or visit the following website:

www.novartisclinicaltrials.com

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-03; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Mean reduction in anxiety from baseline to week 6

SECONDARY OUTCOMES:
The difference on day 4 in effect between placebo and the individual doses of XBD173 on reduction in anxiety and depression
Pharmacokinetic assessments at baseline
Pharmacogenetic assessments at baseline
Pharmacogenomic and proteomic assessments at baseline
Metabonomic assessments at visits 4, 7 and 10

CONTACTS AND LOCATIONS:
Locations (23):
- United States (16):
  - Investigational Site, Anaheim, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Newport Beach, California
  - Investigational Site, Redlands, California
  - Investigational Site, San Diego, California
  - Investigational Site, Fort Meyers, Florida
  - Investigational Site, St. Petersburg, Florida
  - Investigational Site, West Palm Beach, Florida
  - Investigational Site, Atlanta, Georgia
  - Investigational Site, Hoffman Estates, Illinois
  - Investigational Site, Oak Brook, Illinois
  - Investigational Site, Overland Park, Kansas
  - Investigational Site, Dayton, Ohio
  - Investigational Site, Portland, Oregon
  - Investigational Site, Madison, Tennessee
  - Investigational Site, Memphis, Tennessee
- Canada (7):
  - Investigational Site, Edmonton, Alberta
  - Investigational Site, Kelowna, British Columbia
  - Investigational Site, Hamilton, Ontario
  - Investigational Site, Ottawa, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Montreal, Quebec
  - Investigational Site, Sherbrooke, Quebec